CLINICAL TRIAL: NCT00802399
Title: Partial Lacrimal Punctual Occlusion in the Management of Dry Eye
Brief Title: Partial Lacrimal Punctual Occlusion
Acronym: PLPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Ricardo Holzchuh/ MD, Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0300/08
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2008-08

CONDITIONS: Dry Eye
Keywords: Cornea; Dry eye; lacrimal punctual occlusion; lacrimal film; ocular surface
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Partial Lacrimal Punctual Occlusion (Other): Cauterization of the edge of all lacrimal punctum was carried out in all patients
  Interventions: Procedure: Partial Lacrimal Punctual Occlusion

INTERVENTIONS:
Procedure: Partial Lacrimal Punctual Occlusion — Cauterization of the edge of all lacrimal punctum was carried out in all patients

SUMMARY:
The purpose of this study is to describe a case series of patients with chronic dry eye submitted to partial punctual occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Sin and symptom of dry eye
* Use more than 4 times a day topic lubricant for the eye

Exclusion Criteria:

* Ocular diseases other than dry eye
* Use of systemic drugs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Holzchuh, MD, Principal Investigator — Instituto do Coracao
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil